CLINICAL TRIAL: NCT04212936
Title: Optimum-pressure for Reducing Postoperative Shoulder-tip Pain in Laparoscopic Cholecystectomy, a Prospective Randomized Controlled Trial
Brief Title: Optimum-pressure for Reducing Postoperative Shoulder-tip Pain in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Narongsak Rungsakulkij, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2019/1005
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 8 mmHg pressure group
- Study group (Experimental): 10 mmHg group
  Interventions: Procedure: Intraabdominal pressure

INTERVENTIONS:
Procedure: Intraabdominal pressure — Limited intraabdominal pressure during laparoscopic cholecystectomy between 8 and 10 mmHg.
  Arms: Study group

SUMMARY:
Laparoscopic cholecystectomy (LC) is the standard treatment of gallbladder disease. LC is the common procedure for general surgeons. Although LC is a safe procedure with very low mortality (<1%), it has some associated major morbidity. Bile duct injury is the most serious complication of LC. However, there are some postoperative morbidity including shoulder-tip pain. The incidence of shoulder-tip pain is about 15-45%, which might be influencing the patient outcome including length of hospital stay. From the previous studies, one of the important factor associated with this condition is pneumoperitoneum pressure. Thus, the suggestion of the intra-abdominal pressure should be low pressure as about 8 mmHg. However, the optimum pressure for the low-pressure during laparoscopic cholecystectomy is controversial.

DETAILED DESCRIPTION:
We designed the prospective randomized controlled trial to comparing the postoperative shoulder tip pain between two low pressure level (8 and 10 mmHg) during laparoscopic cholecystectomy. After the enrolled participant signed the inform consent, the participant was randomly assigned to 8 or 10 mmHg group. The standard procedure of the laparoscopic cholecystectomy was performed by experience surgeons. During the operation, the pressure limit can be adjusted to facilitate the procedure according to the surgeons. Following the operation, the investigator will ask about the shoulder tip pain from the participant during 48 hours. The standard of care including pain medication during postoperative period was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 15 years
2. Elective procedure of laparoscopic cholecystectomy
3. Sign to Inform consent

Exclusion Criteria:

1. Emergency surgery
2. Concomitant other procedure performed
3. Deny to participant

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-12-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder tip pain | 48 hours
  The shoulder tip pain was assessed by the investigator during postoperative period unfil 48 hours. The measurement of the outcome, the investigator would ask the participant by the clinical record form and questionnair. The answer of the questionnaire is presence or absence of the shoulder pain or pain around the shoulder and scapular region.

SECONDARY OUTCOMES:
Change of intra-abdominal pressure | Immediately after surgery
  The change of intra-abminal pressure was measure by two parameters. Firstly, the adjustment of the pressure during the operation was recorded by the questionnaire. The answer of the questionnaire is the presence or absence of the intra-abdominal pressure change. Secondly, the maximum intra-abdominal pressure which is the highest pressure used during the operation, is measure by the level of the pressure appearing in the laparoscopic station by mmHg unit.
Difficulty of the operation | Immediately after surgery
  The difficulty level of the operation which evaluated by the surgeons. The measurement of this outcome by the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Narongsak Rungsakulkij, M.D., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No